CLINICAL TRIAL: NCT00405678
Title: The Effects of Exercise Training on Tumor Vascularity and Response to Neoadjuvant Therapy in Operable Breast Cancer: A Phase I-II Study
Brief Title: Exercise Intervention Study for Early-Stage Breast Cancer Patients Receiving Neoadjuvant Therapy.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00007112; 8426 (Other: Duke legacy protocol number)
Record Dates: First submitted 2006-11-29; First posted 2006-11-30 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Breast Cancer
Keywords: Exercise Intervention; Breast Cancer; Neo-Adjuvant Therapy; Operable Breast Cancer Stage I-II receiving neo-adjuvant chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Exercise

ARMS (2):
- 1 (Experimental): Subjects receiving chemo and exercise training
  Interventions: Behavioral: Exercise Training
- 2 (Experimental): Subjects receiving chemo only
  Interventions: Behavioral: Exercise Training; Behavioral: Chemo only

INTERVENTIONS:
Behavioral: Exercise Training — Subjects receiving chemo with exercise training
Behavioral: Chemo only — Subjects receiving chemo only
  Arms: 2

SUMMARY:
To determine the effects of endurance exercise training on cardiopulmonary fitness in breast cancer patients undergoing neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
Given that this is the first study to explore the potential effects of exercise training on exercise capacity, tumor vascularity and response in women undergoing neoadjuvant chemotherapy for operable breast cancer, prior to the initiation of the full investigation, we will conduct a small vanguard study to ensure we can achieve acceptable exercise adherence rates in the absence of dose-limiting toxicities (DLTs). Specifically, three operable breast cancer patients will be recruited and enrolled as described below and perform exercise training for a minimum of six weeks. If acceptable exercise rates are observed in the absence of severe DLTs during this time, we will proceed with the full investigation (recruitment of additional 20 patients) (see Figure 2). Using a prospective, randomized design, potential participants will be identified and screened for eligibility by an assigned Breast Protocol Nurse (TBD) via medical record review of patients scheduled for their primary neoadjuvant chemotherapy consultation at DCCC

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed operable primary breast cancer
* Age 18 or older
* Karnofsky performance status greater than 70
* No previous malignancy
* Absence of significant cardiac disease (left ventricular ejection fraction greater than or equal to 50%)
* No hormonal replacement therapy use within the past month
* Not pregnant
* Ability to read and understand English
* Signed written informed consent prior to beginning protocol specific procedures
* Willing to travel to DUMC to exercise three times per week
* Primary treating oncologist approval

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2006-09; Primary Completion 2010-02 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Determine effects of endurance exercise training on cardiopulmonary fitness via a stress test | 3 months

SECONDARY OUTCOMES:
Adherence to fitness program | 3 months
Quality of life as determined by the (Functional Assessment of Cancer Therapy-Breast) FACT-B scale. | 3 months
Determine and define feasibility for an adequately powered Phase III study. | 3 months
Determine effects of exercise training on tumor vascularity, systemic response and tumor response. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Lee W Jones, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] American Cancer Society (2005). Cancer: Facts and Figures. ACS, Atlanta, GA.
- [Background] Cole BF, Gelber RD, Gelber S, Coates AS, Goldhirsch A. Polychemotherapy for early breast cancer: an overview of the randomised clinical trials with quality-adjusted survival analysis. Lancet. 2001 Jul 28;358(9278):277-86. doi: 10.1016/S0140-6736(01)05483-6. PMID 11498214
- [Background] Cutuli B, Fourquet A, Luporsi E, Arnould L, Caron Y, Cremoux Pd, Dilhuydy JM, Fondrinier E, Fourme E, Giard-Lefevre S, Blanc-Onfroy ML, Lemanski C, Mauriac L, Sigal-Zafrani B, Tardivon A, This P, Tunon de Lara C, Kirova Y, Fabre N; Federation of French Cancer Centres (FNCLCC), et le groupe de travail SOR. [Standards, Options and Recommendations for the management of ductal carcinoma in situ of the breast (DCIS): update 2004]. Bull Cancer. 2005 Feb;92(2):155-68. French. PMID 15749645
- [Background] Goldhirsch A, Glick JH, Gelber RD, Coates AS, Senn HJ. Meeting highlights: International Consensus Panel on the Treatment of Primary Breast Cancer. Seventh International Conference on Adjuvant Therapy of Primary Breast Cancer. J Clin Oncol. 2001 Sep 15;19(18):3817-27. doi: 10.1200/JCO.2001.19.18.3817. No abstract available. PMID 11559719
- [Background] Rauschecker H, Clarke M, Gatzemeier W, Recht A. Systemic therapy for treating locoregional recurrence in women with breast cancer. Cochrane Database Syst Rev. 2001;2001(4):CD002195. doi: 10.1002/14651858.CD002195. PMID 11687148
- [Background] Wilcken N, Hornbuckle J, Ghersi D. Chemotherapy alone versus endocrine therapy alone for metastatic breast cancer. Cochrane Database Syst Rev. 2003;2003(2):CD002747. doi: 10.1002/14651858.CD002747. PMID 12804433
- [Background] Curnis F, Sacchi A, Corti A. Improving chemotherapeutic drug penetration in tumors by vascular targeting and barrier alteration. J Clin Invest. 2002 Aug;110(4):475-82. doi: 10.1172/JCI15223. PMID 12189241
- [Background] Sherman-Baust CA, Weeraratna AT, Rangel LB, Pizer ES, Cho KR, Schwartz DR, Shock T, Morin PJ. Remodeling of the extracellular matrix through overexpression of collagen VI contributes to cisplatin resistance in ovarian cancer cells. Cancer Cell. 2003 Apr;3(4):377-86. doi: 10.1016/s1535-6108(03)00058-8. PMID 12726863
- [Background] Tannock IF. Tumor physiology and drug resistance. Cancer Metastasis Rev. 2001;20(1-2):123-32. doi: 10.1023/a:1013125027697. PMID 11831640
- [Background] Tannock IF, Lee CM, Tunggal JK, Cowan DS, Egorin MJ. Limited penetration of anticancer drugs through tumor tissue: a potential cause of resistance of solid tumors to chemotherapy. Clin Cancer Res. 2002 Mar;8(3):878-84. PMID 11895922
- [Background] Au JL, Jang SH, Wientjes MG. Clinical aspects of drug delivery to tumors. J Control Release. 2002 Jan 17;78(1-3):81-95. doi: 10.1016/s0168-3659(01)00488-6. PMID 11772451
- [Background] Izumi Y, Xu L, di Tomaso E, Fukumura D, Jain RK. Tumour biology: herceptin acts as an anti-angiogenic cocktail. Nature. 2002 Mar 21;416(6878):279-80. doi: 10.1038/416279b. PMID 11907566
- [Background] Jain RK. Normalizing tumor vasculature with anti-angiogenic therapy: a new paradigm for combination therapy. Nat Med. 2001 Sep;7(9):987-9. doi: 10.1038/nm0901-987. No abstract available. PMID 11533692
- [Background] Jain RK. Normalization of tumor vasculature: an emerging concept in antiangiogenic therapy. Science. 2005 Jan 7;307(5706):58-62. doi: 10.1126/science.1104819. PMID 15637262
- [Background] Padera TP, Stoll BR, Tooredman JB, Capen D, di Tomaso E, Jain RK. Pathology: cancer cells compress intratumour vessels. Nature. 2004 Feb 19;427(6976):695. doi: 10.1038/427695a. PMID 14973470
- [Background] Tong RT, Boucher Y, Kozin SV, Winkler F, Hicklin DJ, Jain RK. Vascular normalization by vascular endothelial growth factor receptor 2 blockade induces a pressure gradient across the vasculature and improves drug penetration in tumors. Cancer Res. 2004 Jun 1;64(11):3731-6. doi: 10.1158/0008-5472.CAN-04-0074. PMID 15172975
- [Background] Winkler F, Kozin SV, Tong RT, Chae SS, Booth MF, Garkavtsev I, Xu L, Hicklin DJ, Fukumura D, di Tomaso E, Munn LL, Jain RK. Kinetics of vascular normalization by VEGFR2 blockade governs brain tumor response to radiation: role of oxygenation, angiopoietin-1, and matrix metalloproteinases. Cancer Cell. 2004 Dec;6(6):553-63. doi: 10.1016/j.ccr.2004.10.011. PMID 15607960
- [Background] Gruber G, Greiner RH, Hlushchuk R, Aebersold DM, Altermatt HJ, Berclaz G, Djonov V. Hypoxia-inducible factor 1 alpha in high-risk breast cancer: an independent prognostic parameter? Breast Cancer Res. 2004;6(3):R191-8. doi: 10.1186/bcr775. Epub 2004 Mar 9. PMID 15084243
- [Background] van Diest PJ, Vleugel MM, van der Groep P, van der Wall E. VEGF-D and HIF-1alpha in breast cancer. J Clin Pathol. 2005 Mar;58(3):335; author reply 336. No abstract available. PMID 15735177
- [Background] van Diest PJ, Vleugel MM, van der Wall E. Expression of HIF-1alpha in human tumours. J Clin Pathol. 2005 Mar;58(3):335-6. No abstract available. PMID 15735176
- [Background] Vleugel MM, Greijer AE, Shvarts A, van der Groep P, van Berkel M, Aarbodem Y, van Tinteren H, Harris AL, van Diest PJ, van der Wall E. Differential prognostic impact of hypoxia induced and diffuse HIF-1alpha expression in invasive breast cancer. J Clin Pathol. 2005 Feb;58(2):172-7. doi: 10.1136/jcp.2004.019885. PMID 15677538
- [Background] Beasley NJ, Leek R, Alam M, Turley H, Cox GJ, Gatter K, Millard P, Fuggle S, Harris AL. Hypoxia-inducible factors HIF-1alpha and HIF-2alpha in head and neck cancer: relationship to tumor biology and treatment outcome in surgically resected patients. Cancer Res. 2002 May 1;62(9):2493-7. PMID 11980639
- [Background] Erler JT, Cawthorne CJ, Williams KJ, Koritzinsky M, Wouters BG, Wilson C, Miller C, Demonacos C, Stratford IJ, Dive C. Hypoxia-mediated down-regulation of Bid and Bax in tumors occurs via hypoxia-inducible factor 1-dependent and -independent mechanisms and contributes to drug resistance. Mol Cell Biol. 2004 Apr;24(7):2875-89. doi: 10.1128/MCB.24.7.2875-2889.2004. PMID 15024076
- [Background] Frederiksen LJ, Siemens DR, Heaton JP, Maxwell LR, Adams MA, Graham CH. Hypoxia induced resistance to doxorubicin in prostate cancer cells is inhibited by low concentrations of glyceryl trinitrate. J Urol. 2003 Sep;170(3):1003-7. doi: 10.1097/01.ju.0000081126.71235.e0. PMID 12913759
- [Background] Harris AL. Hypoxia--a key regulatory factor in tumour growth. Nat Rev Cancer. 2002 Jan;2(1):38-47. doi: 10.1038/nrc704. PMID 11902584
- [Background] Schindl M, Schoppmann SF, Samonigg H, Hausmaninger H, Kwasny W, Gnant M, Jakesz R, Kubista E, Birner P, Oberhuber G; Austrian Breast and Colorectal Cancer Study Group. Overexpression of hypoxia-inducible factor 1alpha is associated with an unfavorable prognosis in lymph node-positive breast cancer. Clin Cancer Res. 2002 Jun;8(6):1831-7. PMID 12060624
- [Background] Williams KJ, Cowen RL, Stratford IJ. Hypoxia and oxidative stress. Tumour hypoxia--therapeutic considerations. Breast Cancer Res. 2001;3(5):328-31. doi: 10.1186/bcr316. Epub 2001 Aug 7. PMID 11597323
- [Background] Yokoi K, Fidler IJ. Hypoxia increases resistance of human pancreatic cancer cells to apoptosis induced by gemcitabine. Clin Cancer Res. 2004 Apr 1;10(7):2299-306. doi: 10.1158/1078-0432.ccr-03-0488. PMID 15073105
- [Background] Kabbinavar FF, Schulz J, McCleod M, Patel T, Hamm JT, Hecht JR, Mass R, Perrou B, Nelson B, Novotny WF. Addition of bevacizumab to bolus fluorouracil and leucovorin in first-line metastatic colorectal cancer: results of a randomized phase II trial. J Clin Oncol. 2005 Jun 1;23(16):3697-705. doi: 10.1200/JCO.2005.05.112. Epub 2005 Feb 28. PMID 15738537
- [Background] Miller KD, Chap LI, Holmes FA, Cobleigh MA, Marcom PK, Fehrenbacher L, Dickler M, Overmoyer BA, Reimann JD, Sing AP, Langmuir V, Rugo HS. Randomized phase III trial of capecitabine compared with bevacizumab plus capecitabine in patients with previously treated metastatic breast cancer. J Clin Oncol. 2005 Feb 1;23(4):792-9. doi: 10.1200/JCO.2005.05.098. PMID 15681523
- [Background] Hurwitz H, Fehrenbacher L, Novotny W, Cartwright T, Hainsworth J, Heim W, Berlin J, Baron A, Griffing S, Holmgren E, Ferrara N, Fyfe G, Rogers B, Ross R, Kabbinavar F. Bevacizumab plus irinotecan, fluorouracil, and leucovorin for metastatic colorectal cancer. N Engl J Med. 2004 Jun 3;350(23):2335-42. doi: 10.1056/NEJMoa032691. PMID 15175435
- [Background] Edwards DG, Schofield RS, Lennon SL, Pierce GL, Nichols WW, Braith RW. Effect of exercise training on endothelial function in men with coronary artery disease. Am J Cardiol. 2004 Mar 1;93(5):617-20. doi: 10.1016/j.amjcard.2003.11.032. PMID 14996592
- [Background] Fogarty JA, Muller-Delp JM, Delp MD, Mattox ML, Laughlin MH, Parker JL. Exercise training enhances vasodilation responses to vascular endothelial growth factor in porcine coronary arterioles exposed to chronic coronary occlusion. Circulation. 2004 Feb 10;109(5):664-70. doi: 10.1161/01.CIR.0000112580.31594.F9. PMID 14769688
- [Background] Gielen S, Hambrecht R. Effects of exercise training on vascular function and myocardial perfusion. Cardiol Clin. 2001 Aug;19(3):357-68. doi: 10.1016/s0733-8651(05)70222-8. PMID 11570110
- [Background] Green DJ, Maiorana A, O'Driscoll G, Taylor R. Effect of exercise training on endothelium-derived nitric oxide function in humans. J Physiol. 2004 Nov 15;561(Pt 1):1-25. doi: 10.1113/jphysiol.2004.068197. Epub 2004 Sep 16. PMID 15375191
- [Background] Hambrecht R, Adams V, Erbs S, Linke A, Krankel N, Shu Y, Baither Y, Gielen S, Thiele H, Gummert JF, Mohr FW, Schuler G. Regular physical activity improves endothelial function in patients with coronary artery disease by increasing phosphorylation of endothelial nitric oxide synthase. Circulation. 2003 Jul 1;107(25):3152-8. doi: 10.1161/01.CIR.0000074229.93804.5C. Epub 2003 Jun 16. PMID 12810615
- [Background] Hambrecht R, Wolf A, Gielen S, Linke A, Hofer J, Erbs S, Schoene N, Schuler G. Effect of exercise on coronary endothelial function in patients with coronary artery disease. N Engl J Med. 2000 Feb 17;342(7):454-60. doi: 10.1056/NEJM200002173420702. PMID 10675425
- [Background] Kingwell BA. Nitric oxide-mediated metabolic regulation during exercise: effects of training in health and cardiovascular disease. FASEB J. 2000 Sep;14(12):1685-96. doi: 10.1096/fj.99-0896rev. PMID 10973917
- [Background] Kingwell BA. Nitric oxide as a metabolic regulator during exercise: effects of training in health and disease. Clin Exp Pharmacol Physiol. 2000 Apr;27(4):239-50. doi: 10.1046/j.1440-1681.2000.03232.x. PMID 10779120
- [Background] Kingwell BA, Jennings GL, Dart AM. Exercise and endothelial function. Circulation. 2000 Nov 28;102(22):E179. doi: 10.1161/01.cir.102.22.e179. No abstract available. PMID 11094053
- [Background] Allen JD, Geaghan JP, Greenway F, Welsch MA. Time course of improved flow-mediated dilation after short-term exercise training. Med Sci Sports Exerc. 2003 May;35(5):847-53. doi: 10.1249/01.MSS.0000064931.62916.8A. PMID 12750596
- [Background] Allen JD, Welsch M, Aucoin N, Wood R, Lee M, LeBlanc KE. Forearm vasoreactivity in type 1diabetic subjects. Can J Appl Physiol. 2001 Feb;26(1):34-43. doi: 10.1139/h01-003. English, French. PMID 11173668
- [Background] Hambrecht R, Fiehn E, Weigl C, Gielen S, Hamann C, Kaiser R, Yu J, Adams V, Niebauer J, Schuler G. Regular physical exercise corrects endothelial dysfunction and improves exercise capacity in patients with chronic heart failure. Circulation. 1998 Dec 15;98(24):2709-15. doi: 10.1161/01.cir.98.24.2709. PMID 9851957
- [Background] Walsh JH, Bilsborough W, Maiorana A, Best M, O'Driscoll GJ, Taylor RR, Green DJ. Exercise training improves conduit vessel function in patients with coronary artery disease. J Appl Physiol (1985). 2003 Jul;95(1):20-5. doi: 10.1152/japplphysiol.00012.2003. PMID 12794092
- [Background] Adams V, Lenk K, Linke A, Lenz D, Erbs S, Sandri M, Tarnok A, Gielen S, Emmrich F, Schuler G, Hambrecht R. Increase of circulating endothelial progenitor cells in patients with coronary artery disease after exercise-induced ischemia. Arterioscler Thromb Vasc Biol. 2004 Apr;24(4):684-90. doi: 10.1161/01.ATV.0000124104.23702.a0. Epub 2004 Feb 26. PMID 14988094
- [Background] Laufs U, Werner N, Link A, Endres M, Wassmann S, Jurgens K, Miche E, Bohm M, Nickenig G. Physical training increases endothelial progenitor cells, inhibits neointima formation, and enhances angiogenesis. Circulation. 2004 Jan 20;109(2):220-6. doi: 10.1161/01.CIR.0000109141.48980.37. Epub 2003 Dec 22. PMID 14691039
- [Background] Rehman J, Li J, Parvathaneni L, Karlsson G, Panchal VR, Temm CJ, Mahenthiran J, March KL. Exercise acutely increases circulating endothelial progenitor cells and monocyte-/macrophage-derived angiogenic cells. J Am Coll Cardiol. 2004 Jun 16;43(12):2314-8. doi: 10.1016/j.jacc.2004.02.049. PMID 15193699
- [Background] Asahara T, Murohara T, Sullivan A, Silver M, van der Zee R, Li T, Witzenbichler B, Schatteman G, Isner JM. Isolation of putative progenitor endothelial cells for angiogenesis. Science. 1997 Feb 14;275(5302):964-7. doi: 10.1126/science.275.5302.964. PMID 9020076
- [Background] Dimmeler S, Aicher A, Vasa M, Mildner-Rihm C, Adler K, Tiemann M, Rutten H, Fichtlscherer S, Martin H, Zeiher AM. HMG-CoA reductase inhibitors (statins) increase endothelial progenitor cells via the PI 3-kinase/Akt pathway. J Clin Invest. 2001 Aug;108(3):391-7. doi: 10.1172/JCI13152. PMID 11489932
- [Background] Jiang S, Walker L, Afentoulis M, Anderson DA, Jauron-Mills L, Corless CL, Fleming WH. Transplanted human bone marrow contributes to vascular endothelium. Proc Natl Acad Sci U S A. 2004 Nov 30;101(48):16891-6. doi: 10.1073/pnas.0404398101. Epub 2004 Nov 17. PMID 15548607
- [Background] Kalka C, Masuda H, Takahashi T, Kalka-Moll WM, Silver M, Kearney M, Li T, Isner JM, Asahara T. Transplantation of ex vivo expanded endothelial progenitor cells for therapeutic neovascularization. Proc Natl Acad Sci U S A. 2000 Mar 28;97(7):3422-7. doi: 10.1073/pnas.97.7.3422. PMID 10725398
- [Background] Llevadot J, Murasawa S, Kureishi Y, Uchida S, Masuda H, Kawamoto A, Walsh K, Isner JM, Asahara T. HMG-CoA reductase inhibitor mobilizes bone marrow--derived endothelial progenitor cells. J Clin Invest. 2001 Aug;108(3):399-405. doi: 10.1172/JCI13131. PMID 11489933
- [Background] Murohara T, Ikeda H, Duan J, Shintani S, Sasaki Ki, Eguchi H, Onitsuka I, Matsui K, Imaizumi T. Transplanted cord blood-derived endothelial precursor cells augment postnatal neovascularization. J Clin Invest. 2000 Jun;105(11):1527-36. doi: 10.1172/JCI8296. PMID 10841511
- [Background] Takahashi T, Kalka C, Masuda H, Chen D, Silver M, Kearney M, Magner M, Isner JM, Asahara T. Ischemia- and cytokine-induced mobilization of bone marrow-derived endothelial progenitor cells for neovascularization. Nat Med. 1999 Apr;5(4):434-8. doi: 10.1038/7434. PMID 10202935
- [Background] Urbich C, Heeschen C, Aicher A, Sasaki K, Bruhl T, Farhadi MR, Vajkoczy P, Hofmann WK, Peters C, Pennacchio LA, Abolmaali ND, Chavakis E, Reinheckel T, Zeiher AM, Dimmeler S. Cathepsin L is required for endothelial progenitor cell-induced neovascularization. Nat Med. 2005 Feb;11(2):206-13. doi: 10.1038/nm1182. Epub 2005 Jan 23. PMID 15665831
- [Background] Teicher BA. A systems approach to cancer therapy. (Antioncogenics + standard cytotoxics-->mechanism(s) of interaction). Cancer Metastasis Rev. 1996 Jun;15(2):247-72. doi: 10.1007/BF00437479. No abstract available. PMID 8842498
- [Background] Jones LW, Eves ND, Courneya KS, Chiu BK, Baracos VE, Hanson J, Johnson L, Mackey JR. Effects of exercise training on antitumor efficacy of doxorubicin in MDA-MB-231 breast cancer xenografts. Clin Cancer Res. 2005 Sep 15;11(18):6695-8. doi: 10.1158/1078-0432.CCR-05-0844. PMID 16166449
- [Background] Zielinski MR, Muenchow M, Wallig MA, Horn PL, Woods JA. Exercise delays allogeneic tumor growth and reduces intratumoral inflammation and vascularization. J Appl Physiol (1985). 2004 Jun;96(6):2249-56. doi: 10.1152/japplphysiol.01210.2003. Epub 2004 Mar 12. PMID 15020578
- [Background] Courneya KS, Mackey JR, Bell GJ, Jones LW, Field CJ, Fairey AS. Randomized controlled trial of exercise training in postmenopausal breast cancer survivors: cardiopulmonary and quality of life outcomes. J Clin Oncol. 2003 May 1;21(9):1660-8. doi: 10.1200/JCO.2003.04.093. PMID 12721239
- [Background] Blair SN, Kampert JB, Kohl HW 3rd, Barlow CE, Macera CA, Paffenbarger RS Jr, Gibbons LW. Influences of cardiorespiratory fitness and other precursors on cardiovascular disease and all-cause mortality in men and women. JAMA. 1996 Jul 17;276(3):205-10. PMID 8667564
- [Background] Myers J, Prakash M, Froelicher V, Do D, Partington S, Atwood JE. Exercise capacity and mortality among men referred for exercise testing. N Engl J Med. 2002 Mar 14;346(11):793-801. doi: 10.1056/NEJMoa011858. PMID 11893790
- [Background] Jones LW, Courneya KS, Fairey AS, Mackey JR. Does the theory of planned behavior mediate the effects of an oncologist's recommendation to exercise in newly diagnosed breast cancer survivors? Results from a randomized controlled trial. Health Psychol. 2005 Mar;24(2):189-97. doi: 10.1037/0278-6133.24.2.189. PMID 15755233
- [Background] Jones LW, Courneya KS, Fairey AS, Mackey JR. Effects of an oncologist's recommendation to exercise on self-reported exercise behavior in newly diagnosed breast cancer survivors: a single-blind, randomized controlled trial. Ann Behav Med. 2004 Oct;28(2):105-13. doi: 10.1207/s15324796abm2802_5. PMID 15454357
- [Background] Jones LW, Courneya KS. Exercise counseling and programming preferences of cancer survivors. Cancer Pract. 2002 Jul-Aug;10(4):208-15. doi: 10.1046/j.1523-5394.2002.104003.x. PMID 12100105
- [Background] Jones LW, Courneya KS. Exercise discussions during cancer treatment consultations. Cancer Pract. 2002 Mar-Apr;10(2):66-74. doi: 10.1046/j.1523-5394.2002.102004.x. PMID 11903271
- [Background] Segal RJ, Reid RD, Courneya KS, Malone SC, Parliament MB, Scott CG, Venner PM, Quinney HA, Jones LW, D'Angelo ME, Wells GA. Resistance exercise in men receiving androgen deprivation therapy for prostate cancer. J Clin Oncol. 2003 May 1;21(9):1653-9. doi: 10.1200/JCO.2003.09.534. PMID 12721238
- [Background] Therasse P, Arbuck SG, Eisenhauer EA, Wanders J, Kaplan RS, Rubinstein L, Verweij J, Van Glabbeke M, van Oosterom AT, Christian MC, Gwyther SG. New guidelines to evaluate the response to treatment in solid tumors. European Organization for Research and Treatment of Cancer, National Cancer Institute of the United States, National Cancer Institute of Canada. J Natl Cancer Inst. 2000 Feb 2;92(3):205-16. doi: 10.1093/jnci/92.3.205. PMID 10655437
- [Background] Verma S, Anderson TJ. Fundamentals of endothelial function for the clinical cardiologist. Circulation. 2002 Feb 5;105(5):546-9. doi: 10.1161/hc0502.104540. No abstract available. PMID 11827916
- [Background] Zhang ZG, Zhang L, Jiang Q, Chopp M. Bone marrow-derived endothelial progenitor cells participate in cerebral neovascularization after focal cerebral ischemia in the adult mouse. Circ Res. 2002 Feb 22;90(3):284-8. doi: 10.1161/hh0302.104460. PMID 11861416
- [Background] Allen JD, Cobb FR, Gow AJ. Regional and whole-body markers of nitric oxide production following hyperemic stimuli. Free Radic Biol Med. 2005 May 1;38(9):1164-9. doi: 10.1016/j.freeradbiomed.2004.12.018. PMID 15808413
- [Background] Brady MJ, Cella DF, Mo F, Bonomi AE, Tulsky DS, Lloyd SR, Deasy S, Cobleigh M, Shiomoto G. Reliability and validity of the Functional Assessment of Cancer Therapy-Breast quality-of-life instrument. J Clin Oncol. 1997 Mar;15(3):974-86. doi: 10.1200/JCO.1997.15.3.974. PMID 9060536
- [Background] Cella D. The Functional Assessment of Cancer Therapy-Anemia (FACT-An) Scale: a new tool for the assessment of outcomes in cancer anemia and fatigue. Semin Hematol. 1997 Jul;34(3 Suppl 2):13-9. PMID 9253779
- [Background] Stables GJ, Subar AF, Patterson BH, Dodd K, Heimendinger J, Van Duyn MA, Nebeling L. Changes in vegetable and fruit consumption and awareness among US adults: results of the 1991 and 1997 5 A Day for Better Health Program surveys. J Am Diet Assoc. 2002 Jun;102(6):809-17. doi: 10.1016/s0002-8223(02)90181-1. PMID 12067046
- [Background] Demark-Wahnefried W, Clipp EC, McBride C, Lobach DF, Lipkus I, Peterson B, Clutter Snyder D, Sloane R, Arbanas J, Kraus WE. Design of FRESH START: a randomized trial of exercise and diet among cancer survivors. Med Sci Sports Exerc. 2003 Mar;35(3):415-24. doi: 10.1249/01.MSS.0000053704.28156.0F. PMID 12618570
- [Background] Demark-Wahnefried W, Morey MC, Clipp EC, Pieper CF, Snyder DC, Sloane R, Cohen HJ. Leading the Way in Exercise and Diet (Project LEAD): intervening to improve function among older breast and prostate cancer survivors. Control Clin Trials. 2003 Apr;24(2):206-23. doi: 10.1016/s0197-2456(02)00266-0. PMID 12689742
- [Background] Godin G, Jobin J, Bouillon J. Assessment of leisure time exercise behavior by self-report: a concurrent validity study. Can J Public Health. 1986 Sep-Oct;77(5):359-62. No abstract available. PMID 3791117
- [Background] Godin G, Shephard RJ. A simple method to assess exercise behavior in the community. Can J Appl Sport Sci. 1985 Sep;10(3):141-6. PMID 4053261
- [Background] Segal R, Evans W, Johnson D, Smith J, Colletta S, Gayton J, Woodard S, Wells G, Reid R. Structured exercise improves physical functioning in women with stages I and II breast cancer: results of a randomized controlled trial. J Clin Oncol. 2001 Feb 1;19(3):657-65. doi: 10.1200/JCO.2001.19.3.657. PMID 11157015